CLINICAL TRIAL: NCT00383279
Title: Improving Employment Among Gynecologic Cancer Survivors
Brief Title: Improving Employment in Patients Who Have Survived Cervical Cancer, Uterine Cancer, or Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Other
Other Study IDs: CCCWFU-99106; CCCWFU-99106; CCCWFU-BG06-014
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Cervical Cancer; Ovarian Cancer; Sarcoma
Keywords: recurrent cervical cancer; stage 0 cervical cancer; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; recurrent uterine sarcoma; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; ovarian stromal cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage I ovarian epithelial cancer; stage I ovarian germ cell tumor; stage II ovarian epithelial cancer; stage II ovarian germ cell tumor; stage III ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Sarcoma; Uterine Cervical Dysplasia; Carcinoma, Ovarian Epithelial | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: counseling intervention
Other: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Finding out which problems affect employment in survivors of gynecologic cancer may help in planning cancer treatment and improve the quality of life of future cancer survivors.

PURPOSE: This research study is looking at ways to improve employment in patients who have survived cervical cancer, uterine cancer, or ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Conduct formative work, including 4 to 5 focus groups, leading to development of a structured interview instrument assessing factors related to employment outcomes among women with gynecologic cancers.
* Pilot a recruitment strategy and administer the interview among a sample of 60 to 70 gynecologic cancer survivors; and, with each woman's permission, a family member, a key health care provider, and her supervisor will be interviewed.

OUTLINE: This is a multicenter, pilot study.

Patients complete a survey, meet with a focus group, and undergo a short interview. Patient-designated participants are also interviewed; these individuals may include a health care provider, a significant other, and/or a work supervisor.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following invasive cancers:

  * Cervical cancer
  * Uterine cancer
  * Ovarian cancer
* Diagnosed ≥ 6 months ago
* Any stage disease
* Employed at the time of diagnosis, defined as working for pay ≥ 20 hours/week

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-02 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Development of a structured interview instrument
Recruitment strategy

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte E. Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States